CLINICAL TRIAL: NCT04023526
Title: A Phase 2 Study of Cusatuzumab Plus Azacitidine in Patients With Newly Diagnosed Acute Myeloid Leukemia Who Are Not Candidates for Intensive Chemotherapy
Brief Title: A Study of Cusatuzumab Plus Azacitidine in Participants With Newly Diagnosed Acute Myeloid Leukemia Who Are Not Candidates for Intensive Chemotherapy
Acronym: CULMINATE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OncoVerity, Inc. (Industry)
Collaborators: argenx (Industry); Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CULM20236; 2019-000473-23 (EudraCT Number); CULM20236 (Other: OncoVerity, Inc.); 74494550AML2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-07-16; First posted 2019-07-17 (Actual); Results first posted 2024-07-30 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Azacitidine 75 mg/m^2 and Cusatuzumab 10 mg/kg (Experimental): Participants will receive azacitidine 75 milligram per meter square (mg/m^2) subcutaneously (SC) or intravenously (IV) on Day 1 through Day 7 and cusatuzumab 10 milligram per kilogram (mg/kg) IV on Day 3 and Day 17 of each 28-day cycle in Part 1. Part 1 findings will be reviewed by a data review committee.
  Interventions: Drug: Azacitidine; Drug: Cusatuzumab
- Azacitidine 75 mg/m^2 and Cusatuzumab 20 mg/kg (Experimental): Participants will receive azacitidine 75 mg/m^2 SC or IV on Day 1 through Day 7 and cusatuzumab 20 mg/kg IV on Day 3 and Day 17 of each 28-day cycle in Part 1. Part 1 findings will be reviewed by a data review committee.
  Interventions: Drug: Azacitidine; Drug: Cusatuzumab

INTERVENTIONS:
Drug: Azacitidine — Azacitidine SC or IV will be administered at a standard dose of 75 mg/m^2 on days 1-7 of each cycle.
Drug: Cusatuzumab — Cusatuzumab IV will be administered as 10 mg/kg or 20 mg/kg on days 3 and 17 of each cycle.
  Other Names: OV-1001; JNJ-74494550; ARGX-110

SUMMARY:
The purpose of this study is to determine the efficacy of cusatuzumab in combination with azacitidine in participants with previously untreated acute myeloid leukemia (AML) who are not eligible for intensive chemotherapy.

DETAILED DESCRIPTION:
AML is a heterogeneous disease characterized by uncontrolled clonal expansion of hematopoietic progenitor cells. As the most common form of acute leukemia, AML accounts for the largest number of annual deaths from leukemia. Over 95 percent (%) of AML blasts harvested from newly diagnosed AML participants expressed Cluster of Differentiation (CD) 70 on the cell surface. Cusatuzumab (JNJ-74494550) is a humanized monoclonal antibody of camelid origin, binding with tight affinity to human CD70. Cusatuzumab has been modified to induce enhanced antibody-dependent cell-mediated cytotoxicity (ADCC) for therapeutic use in participants with cancer. Azacitidine is a pyrimidine nucleoside analogue of cytidine with antineoplastic activity and is indicated for the treatment of adult participants with AML or intermediate 2 and high-risk myelodysplastic syndrome (MDS) with greater than 20% marrow blasts who are not eligible for hematopoietic stem cell transplantation. This study will evaluate 2 doses of cusatuzumab in combination with standard dose azacitidine in participants with AML who are not candidates for intensive chemotherapy (Part 1). Part 1 data will be reviewed by a Data Review Committee to select a preferred dose of cusatuzumab. The study will include a Screening Phase (28 days prior to randomization), a Treatment Phase, and a Follow-up Phase. The study includes evaluations like vital signs, electrocardiogram, spirometry test, serum chemistry and hematology tests.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia (AML) according to World Health Organisation (WHO) 2016 criteria and fulfilling all of the following criteria that defines those who are "not candidates for intensive chemotherapy":

  1. greater than or equal to (>=)75 years of age or
  2. less than (<) 75 years of age with at least one of the following comorbidities: Eastern Cooperative Oncology Group (ECOG) Performance Status of 2; Severe cardiac comorbidity defined as congestive heart failure or ejection fraction less than or equal to (<=) 50 percent (%); Severe pulmonary comorbidity defined as documented pulmonary disease with lung diffusing capacity for carbon monoxide (DLCO) <=65% of expected, or forced expiratory volume in 1 second (FEV1) <=65% of expected or dyspnea at rest requiring oxygen; Moderate hepatic impairment defined according to NCI organ dysfunction classification criteria (total bilirubin >=1.5 up to 3 times upper limit of normal [ULN]); Creatinine clearance <45 milliliter per minute per 1.73 meter square (mL/ min/1.73 m^2); Comorbidity that, in the Investigator's opinion, makes the participant unsuitable for intensive chemotherapy and must be documented and approved by the Sponsor before randomization
* De novo or secondary AML
* Previously untreated AML (except: emergency leukapheresis, hydroxyurea, and/or 1 dose of cytarabine [example: 1-2 gram per meter square {g/m^2}] during the Screening Phase to control hyperleukocytosis. These treatments must be discontinued >=24 hours prior to start of study drug). Empiric all trans retinoic acid (ATRA) treatment for presumed acute promyelocytic leukemia (APL) is permitted but APL must be ruled out and ATRA must be discontinued >=24 hours prior to the start of study drug
* Not eligible for an allogeneic hematopoietic stem cell transplantation
* ECOG Performance Status score of 0, 1 or 2

Exclusion Criteria:

* Acute promyelocytic leukemia
* Leukemic involvement or clinical symptoms of leukemic involvement of the central nervous system
* Use of immune suppressive agents for the past 4 weeks before the first administration of cusatuzumab on Cycle 1 Day 3. For regular use of systemic corticosteroids, participants may only be included if free of systemic corticosteroids for a minimum of 5 days before the first administration of cusatuzumab. Treatment of adrenal insufficiency with physiologic replacement doses of corticosteroids are allowed
* Prior treatment with a hypomethylating agent for treatment of AML or myelodysplastic syndrome (MDS)
* Active malignancies (that is, progressing or requiring treatment in the last 24 months) other than the disease being treated under the study
* Any active systemic infection
* Known allergies, hypersensitivity, or intolerance to cusatuzumab or azacitidine or its excipients (that is, mannitol, an excipient of azacitidine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2026-05-15 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clayton Smith, MD, Study Director — OncoVerity, Inc.
Locations (56):
- Australia (5):
  - St Vincents Hospital Sydney, Darlinghurst
  - St Vincents Hospital Melbourne, Fitzroy
  - The Alfred Hospital, Melbourne
  - Royal Perth Hospital, Perth
  - Westmead Hospital, Westmead
- Brazil (2):
  - Universidade Estadual De Campinas, Campinas
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
- France (7):
  - CHU d'Angers, Angers
  - CHU Grenoble, Grenoble
  - Institut Paoli Calmettes, Marseille
  - Centre Hospitalier Universitaire (CHU) de Bordeaux Hopital HautLeveque Centre Francois Magendie, Pessac
  - CHU Lyon Sud, Pierre-Bénite
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
  - CHRU Tours Hôpital Bretonneau, Tours
- Israel (3):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (7):
  - Azienda Opedaliero-Universitaria Policlinico Sant'orsola Malpighi di Bologna, Bologna
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Istituto Europeo di Oncologia, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Division of Hematology, Cardarelli Hospital, Napoli
  - Azienda Sanitaria Universitaria Integrata di Udine, Udine
- Russia (11):
  - Chelyabinck Regional Clinical Hospital, Chelyabinsk
  - S.P. Botkin Moscow City Clinical Hospital, Moscow
  - City Clinical Hospital # 40, Moscow
  - Nizhniy Novgorod Region Clinical Hospital, Nizhny Novgorod
  - Ryazan Regional Clinical Hospital, Ryazan
  - St.-Petersburg Clinical Research Institute of Hematology and Transfusiology, Saint Petersburg
  - City clinical hospital #15, Saint Petersburg
  - Samara Region Clinical Hospital, Samara
  - Oncologic Dispensary No.2, Sochi
  - Komi Republic Oncology dispensary, Syktyvkar
  - Ekaterinburg City Clinical Hospital # 7, Yekaterinburg
- Spain (10):
  - Hosp. Quiron Madrid Pozuelo, Pozuelo de Alarcón, Madrid
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Inst. Cat. Doncologia-H Duran I Reynals, Barcelona
  - Hosp. Univ. Vall D Hebron, Barcelona
  - Hosp. Reina Sofia, Córdoba
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. Son Espases, Palma
  - Hosp. Clinico Univ. de Salamanca, Salamanca
  - Hosp. Univ. I Politecni La Fe, Valencia
- Switzerland (4):
  - Kantonsspital Aarau, Aarau
  - INSELSPITAL, Universitätsspital Bern, Bern
  - Hopitaux Universitaires de Geneve, Geneva
  - UniversitaetsSpital Zuerich, Zurich
- Turkey (Türkiye) (7):
  - Gulhane Egitim ve Arastirma Hastanesi, Ankara
  - Dr.Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara
  - Ankara University Medical Faculty Hematology Department - Hematology, Ankara
  - Istanbul Egitim ve Arastirma Hastanesi, Istanbul
  - Dokuz Eylul Universitesi Tip Fakultesi, Izmir
  - Ondokuz Mayis Universitesi Tip Fakultesi, Samsun
  - Karadeniz Teknik University Medical Faculty, Trabzon

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Pabst T, Papayannidis C, Demirkan F, Doronin V, Fogliatto LM, Guttke C, Gyan E, Hamad N, Herrera P, Hultberg A, Jacobs J, Johnson AJ, Langlois A, Ma X, Martinelli G, Arnan M, Muller R, Nottage K, Ofran Y, Ozcan M, Samoilova O, Tolbert JA, Trudel GC, Xiu L, Vey N, Wei AH. Cusatuzumab plus azacitidine in newly diagnosed acute myeloid leukaemia ineligible for intensive chemotherapy (CULMINATE): part one of a randomised, phase 2, dose optimisation study. Lancet Haematol. 2023 Nov;10(11):e902-e912. doi: 10.1016/S2352-3026(23)00207-7. PMID 37914483

RESULTS

PARTICIPANT FLOW:
Groups:
- Cusatuzumab 10 mg/kg Plus Azacitidine: Participants received azacitidine 75 milligram per meter square (mg/m^2) subcutaneously (SC) or intravenously (IV) on Day 1 through Day 7 and cusatuzumab 10 milligram per kilogram (mg/kg) IV on Day 3 and Day 17 of each 28-day cycle.
- Cusatuzumab 20 mg/kg Plus Azacitidine: Participants received azacitidine 75 mg/m^2 SC or IV on Day 1 through Day 7 and cusatuzumab 20 mg/kg IV on Day 3 and Day 17 of each 28-day cycle.
Period: Overall Study
Arm/Group | Cusatuzumab 10 mg/kg Plus Azacitidine | Cusatuzumab 20 mg/kg Plus Azacitidine
Started | 51 | 52
Completed | 46 | 42
Not Completed | 5 | 10
Not completed — Ongoing treatment at data cutoff | 5 | 9
Not completed — Randomized but did not receive assigned treatment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cusatuzumab 10 mg/kg Plus Azacitidine | Cusatuzumab 20 mg/kg Plus Azacitidine | Total
Number analyzed (Participants) | 51 | 52 | 103
Age, Continuous [Median (Full Range); unit: years] | 74 [54 to 88] | 75 [59 to 88] | 74 [54 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 28 | 29 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 40 | 38 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 14 | 24
Region of Enrollment [Count of Participants; unit: Participants] — Count of Participants
  Participants
    Turkey | 10 | 8 | 18
    Italy | 5 | 3 | 8
    France | 9 | 10 | 19
    Australia | 5 | 4 | 9
    Switzerland | 4 | 4 | 8
    Russia | 13 | 16 | 29
    Spain | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Remission (CR)
Description: Complete remission based on European Leukemia Network (ELN) 2017 response criteria. Defined as bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absences of extramedullary disease; ANC >= 1.0 x10^9/L; platelet count >=100 x 10^9/L
Time Frame: Up to 3 years and 5 months
Population: Intention-to-treat (ITT)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cusatuzumab 10 mg/kg Plus Azacitidine | Cusatuzumab 20 mg/kg Plus Azacitidine
Number analyzed (Participants) | 51 | 52
percentage of participants | 11.76 [5.5 to 23.4] | 26.92 [16.8 to 40.3]

2. Secondary Outcome: Percentage of Participants With CR With Partial Hematological Recovery (CRh)
Description: CRh defined as meeting all criteria for CR except ANC >0.5x10^9/L and platelet count >50x10^9/L
Time Frame: Up to 3 years and 5 months
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cusatuzumab 10 mg/kg Plus Azacitidine | Cusatuzumab 20 mg/kg Plus Azacitidine
Number analyzed (Participants) | 51 | 52
percentage of participants | 9.8 [4.3 to 21] | 7.7 [3 to 18.2]

3. Secondary Outcome: Percentage of Participants With CR Plus CRh
Description: CR plus CRh based on ELN 2017 response criteria. CR defined as bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absences of extramedullary disease; ANC >= 1.0 x10^9/L; platelet count >=100 x 10^9/L CRh defined as meeting all criteria for CR except ANC >0.5x10^9/L and platelet count >50x10^9/L
Time Frame: Up to 3 years and 5 months
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cusatuzumab 10 mg/kg Plus Azacitidine | Cusatuzumab 20 mg/kg Plus Azacitidine
Number analyzed (Participants) | 51 | 52
percentage of participants | 21.6 [12.5 to 34.6] | 34.6 [23.2 to 48.2]

4. Secondary Outcome: Percentage of Participants With CR With Incomplete Recovery (CRi)
Description: CRi based on ELN 2017 response criteria. Defined as meeting all CR criteria except for residual neutropenia (ANC <1.0x10^9/L) or thrombocytopenia (platelets <100x10^9/L)
Time Frame: Up to 3 years and 5 months
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cusatuzumab 20 mg/kg Plus Azacitidine: Participants will received azacitidine 75 mg/m^2 SC or IV on Day 1 through Day 7 and cusatuzumab 20 mg/kg IV on Day 3 and Day 17 of each 28-day cycle.
Arm/Group | Cusatuzumab 10 mg/kg Plus Azacitidine | Cusatuzumab 20 mg/kg Plus Azacitidine
Number analyzed (Participants) | 51 | 52
percentage of participants | 7.8 [3.1 to 18.15] | 5.8 [2 to 15.6]

5. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as percentage of participants with CR, CRh and CRi based on ELN 2017 response criteria.
Time Frame: Up to 3 years and 5 months
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cusatuzumab 10 mg/kg Plus Azacitidine | Cusatuzumab 20 mg/kg Plus Azacitidine
Number analyzed (Participants) | 51 | 52
percentage of participants | 29.4 [18.7 to 43] | 40.4 [28.2 to 53.9]

6. Secondary Outcome: Percentage of Participants With CR Without MRD
Description: CR without minimal residual disease (MRD) defined as less than 1 blast or leukemic stem cell in 1,000 leukocytes (MRD level <10^-3 by flow cytometry).
Time Frame: Up to 3 years and 5 months
Population: ITT
Measure: Count of Participants; unit: Participants
Groups:
- Cusatuzumab 20 mg/kg Plus Azacitidine: Participants will receive azacitidine 75 mg/m^2 SC or IV on Day 1 through Day 7 and cusatuzumab 20 mg/kg IV on Day 3 and Day 17 of each 28-day cycle.
Arm/Group | Cusatuzumab 10 mg/kg Plus Azacitidine | Cusatuzumab 20 mg/kg Plus Azacitidine
Number analyzed (Participants) | 51 | 52
Participants | 1 | 4

7. Secondary Outcome: Percentage of Participants With Negative MRD Who Achieved CR, CRh, CRi, or Morphologic Leukemia-free State (MLFS)
Description: Percentage of participants with negative MRD who achieved CR, CRh, CRi, or MLFS will be reported and is defined as less than (<) 1 blast or leukemic stem cell in 1,000 leukocytes (MRD level <10^-3).
Time Frame: Up to 3 years and 5 months
Reporting Status: Not Posted

8. Secondary Outcome: Time to First Response
Description: Defined as time from randomization to achieving the first response of CR, CRh, or CRi.
Time Frame: Up to 3 years and 5 months
Population: Responder population: Participants who achieved CR, CRh or CRi
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Cusatuzumab 10 mg/kg and Azacitidine: Participants received azacitidine 75 milligram per meter square (mg/m^2) subcutaneously (SC) or intravenously (IV) on Day 1 through Day 7 and cusatuzumab 10 milligram per kilogram (mg/kg) IV on Day 3 and Day 17 of each 28-day cycle.
- Cusatuzumab 20 mg/kg and Azacitidine: Participants received azacitidine 75 mg/m^2 SC or IV on Day 1 through Day 7 and cusatuzumab 20 mg/kg IV on Day 3 and Day 17 of each 28-day cycle.
Arm/Group | Cusatuzumab 10 mg/kg and Azacitidine | Cusatuzumab 20 mg/kg and Azacitidine
Number analyzed (Participants) | 15 | 21
Months | 2.8 [2.6 to 3.5] | 3 [2.8 to 3.9]

9. Secondary Outcome: Duration of First Response
Description: Defined as time from achieving the first response of CR, CRh, or CRi to disease relapse or death from any cause.
Time Frame: Up to 3 years and 5 months
Population: Responder population: Participants who achieved CR, CRh or CRi
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cusatuzumab 10 mg/kg Plus Azacitidine | Cusatuzumab 20 mg/kg Plus Azacitidine
Number analyzed (Participants) | 15 | 21
Months | 5.6 [0.7 to NA] — Upper limit of 95% CI is not estimable due to some participants still being in CR | 13.6 [6.3 to NA] — Upper limit of 95% CI is not estimable due to some participants still being in CR

10. Secondary Outcome: Red Blood Cell (RBC) and/or Platelets Transfusion Independence
Description: Defined as a period of at least 56 consecutive days with no transfusion of RBC and/or platelets between first dose of study drug and the last dose of study drug +30 days.
Time Frame: Up to 3 years and 5 months
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cusatuzumab 10 mg/kg Plus Azacitidine | Cusatuzumab 20 mg/kg Plus Azacitidine
Number analyzed (Participants) | 51 | 52
percentage of participants
  RBC Transfusion Independence | 29.4 [17.5 to 43.8] | 42.3 [28.7 to 56.8]
  Platelets Transfusion Independence | 39.2 [25.8 to 53.9] | 51.9 [37.6 to 66]
  RBC and Platelets Transfusion Independence | 27.5 [15.9 to 41.7] | 36.5 [23.6 to 51]

11. Secondary Outcome: Cusatuzumab Minimum Serum Concentration (Cmin)
Description: Cmin is the minimum cusatuzumab serum concentration observed at Cycle 1 Day 3
Time Frame: Cycle 1 Day 3
Population: All participants with available serum concentrations per intervention group.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter
Arm/Group | Cusatuzumab 10 mg/kg and Azacitidine | Cusatuzumab 20 mg/kg and Azacitidine
Number analyzed (Participants) | 30 | 27
micrograms/milliliter | NA (NA) — Level below the quantification limit | NA (NA) — Level below the quantification limit

12. Secondary Outcome: Maximum Serum Concentration (Cmax) of Cusatuzumab
Description: Cmax is the maximum cusatuzumab serum concentration observed at Cycle 1 Day 3.
Time Frame: Cycle 1 Day 3
Population: All participants with available serum concentrations per intervention group
Measure: Mean (Standard Deviation); unit: micrograms/milliliter
Groups:
- Cusatuzumab 20 mg/kg and Azacitidine: Participants will receive azacitidine 75 mg/m^2 SC or IV on Day 1 through Day 7 and cusatuzumab 20 mg/kg IV on Day 3 and Day 17 of each 28-day cycle.
Arm/Group | Cusatuzumab 10 mg/kg and Azacitidine | Cusatuzumab 20 mg/kg and Azacitidine
Number analyzed (Participants) | 27 | 25
micrograms/milliliter | 224 (54.1) | 458 (89.7)

13. Secondary Outcome: Number of Participants With Anti-cusatuzumab Antibodies
Description: Number of participants exhibiting anti-drug antibodies for cusatuzumab.
Time Frame: Up to 3 years and 5 months
Population: Participants with evaluable samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Cusatuzumab 10 mg/kg Plus Azacitidine | Cusatuzumab 20 mg/kg Plus Azacitidine
Number analyzed (Participants) | 47 | 46
Participants | 7 | 2

ADVERSE EVENTS:
Time Frame: From first dose of study treatment at study day 1 until 30 days after the last dose of study intervention or until the start of subsequent anti-AML therapy (up to approximately 3 years and 5 months)
Description: Treatment emergent events with onset during the intervention phase or that are a consequence of a pre-existing condition that has worsened since baseline.
Groups:
- Cusatuzumab 10 mg/kg Plus Azacitdine: Participants received azacitidine 75 milligram per meter square (mg/m^2) subcutaneously (SC) or intravenously (IV) on Day 1 through Day 7 and cusatuzumab 10 milligram per kilogram (mg/kg) IV on Day 3 and Day 17 of each 28-day cycle.
  .
Arm/Group | Cusatuzumab 10 mg/kg Plus Azacitdine | Cusatuzumab 20 mg/kg Plus Azacitidine
All-Cause Mortality (participants affected / at risk) | 39/51 | 30/51
Serious Adverse Events (participants affected / at risk) | 44/51 | 40/51
Other Adverse Events (participants affected / at risk) | 51/51 | 50/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cusatuzumab 10 mg/kg Plus Azacitdine (N=51) | Cusatuzumab 20 mg/kg Plus Azacitidine (N=51)
Pneumonia (Infections and infestations) | 10 | 9
COVID-19 pneumonia (Infections and infestations) | 2 | 6
Sepsis (Infections and infestations) | 2 | 3
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 2
Septic Shock (Infections and infestations) | 2 | 1
Soft tissue infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 2
COVID-19 (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Pseudomonal sepsis (Infections and infestations) | 1 | 1
Alpha haemolytic streptococcal infection (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Disseminated varicella zoster virus infection (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Injection site abscess (Infections and infestations) | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 1 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Toxic shock syndrome (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Vascular device infection (Infections and infestations) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 10 | 4
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 3
General physical health deterioration (Gastrointestinal disorders) | 2 | 2
Multiple organ dysfunction syndrome (General disorders) | 2 | 2
Sudden death (General disorders) | 3 | 0
Asthenia (General disorders) | 0 | 1
Death (General disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2
Anal fistula (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 2
Renal failure (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Phlebitis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
Cerebral haematoma (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Differentiation syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cusatuzumab 10 mg/kg Plus Azacitdine (N=51) | Cusatuzumab 20 mg/kg Plus Azacitidine (N=51)
Thrombocytopenia (Blood and lymphatic system disorders) | 26 | 30
Anaemia (Blood and lymphatic system disorders) | 24 | 18
Neutropenia (Blood and lymphatic system disorders) | 20 | 21
Leukopenia (Blood and lymphatic system disorders) | 13 | 16
Febrile neutropenia (Blood and lymphatic system disorders) | 11 | 9
Lymphopenia (Blood and lymphatic system disorders) | 13 | 7
Pneumonia (Infections and infestations) | 15 | 13
COVID-19 pneumonia (Infections and infestations) | 2 | 6
Urinary tract infection (Infections and infestations) | 5 | 3
Oral herpes (Infections and infestations) | 3 | 3
Sepsis (Infections and infestations) | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 4 | 1
Diverticulitis (Infections and infestations) | 3 | 0
Oral candidiasis (Infections and infestations) | 0 | 3
Pharyngitis (Infections and infestations) | 0 | 3
Constipation (Gastrointestinal disorders) | 19 | 19
Nausea (Gastrointestinal disorders) | 17 | 19
Diarrhoea (Gastrointestinal disorders) | 15 | 14
Vomiting (Gastrointestinal disorders) | 9 | 11
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Haemorrhoids (Gastrointestinal disorders) | 0 | 5
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Stomatitis (Gastrointestinal disorders) | 3 | 1
Pyrexia (General disorders) | 16 | 15
Asthenia (General disorders) | 8 | 11
Oedema peripheral (General disorders) | 8 | 6
Chills (General disorders) | 3 | 4
Fatigue (General disorders) | 3 | 3
General physical health deterioration (General disorders) | 2 | 3
Hyperthermia (General disorders) | 3 | 0
Non-cardiac chest pain (General disorders) | 0 | 3
Sudden death (General disorders) | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 14 | 8
Decreased appetite (Metabolism and nutrition disorders) | 9 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 9
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Erythema (Skin and subcutaneous tissue disorders) | 5 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Hypotension (Vascular disorders) | 4 | 10
Haematoma (Vascular disorders) | 3 | 6
Hypertension (Vascular disorders) | 2 | 3
Weight decreased (Investigations) | 10 | 7
Alanine aminotransferase increased (Investigations) | 6 | 5
Aspartate aminotransferase increased (Investigations) | 4 | 4
Gamma-glutamyltransferase increased (Investigations) | 1 | 5
Blood alkaline phosphatase increased (Investigations) | 1 | 4
Headache (Nervous system disorders) | 5 | 6
Dizziness (Nervous system disorders) | 1 | 5
Atrial fibrillation (Cardiac disorders) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 5 | 4
Insomnia (Psychiatric disorders) | 2 | 4
Delirium (Psychiatric disorders) | 3 | 0
Renal failure (Renal and urinary disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/26/NCT04023526/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT04023526/SAP_001.pdf